CLINICAL TRIAL: NCT05863416
Title: Adjunctive Dexmedetomidine Infusion in Non-intubated Video-assisted Thoracoscopic Surgery
Brief Title: Dexmedetomidine in Non-intubated VATS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Wei-Cheng Tseng, Principal Investigator, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B202305049_V2
Record Dates: First submitted 2023-05-03; First posted 2023-05-18 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-04

CONDITIONS: Dexmedetomidine; Thoracoscopy; Analgesia
Keywords: Dexmedetomidine; Thoracoscopy; Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Saline (Active Comparator): Propofol-based total intravenous anesthesia with saline infusion
  Interventions: Drug: Dexmedetomidine infusion
- Group Dexmedetomidine (Experimental): Propofol-based total intravenous anesthesia with dexmedetomidine infusion
  Interventions: Drug: Dexmedetomidine infusion

INTERVENTIONS:
Drug: Dexmedetomidine infusion — Intraoperative dexmedetomidine infusion

SUMMARY:
This prospective study aims to evaluate the effectiveness of intraoperative DEX for postoperative analgesia and recovery after non-intubated VATS. In addition, the investigators observe the impact of DEX on anesthetic requirements, hemodynamic parameters, and adverse events during non-intubated VATS.

DETAILED DESCRIPTION:
The non-intubated thoracoscopic approach has been adapted for use with major lung resections. The non-intubated VATS tries to minimize the adverse effects of tracheal intubation and general anesthesia, such as intubation-related airway trauma, ventilation-induced lung injury, residual neuromuscular blockade, and postoperative nausea and vomiting. An adequate analgesia allows VATS to be performed in sedated patients and the potential adverse effects related to general anesthesia and selective ventilation can be avoided. Dexmedetomidine (DEX), a highly selective alpha-2 receptor agonist, is increasingly used in anesthesia with sedative, hypnotic, anxiolytic, sympatholytic, and analgesic effects. It can also attenuate perioperative stress and inflammation and preserve the immunity of surgical patients, which may contribute to reduced postoperative complications and improved clinical outcomes. This study aims to evaluate the effectiveness of intraoperative DEX for postoperative analgesia and recovery after non-intubated VATS. In addition, the investigators observe the impact of DEX on anesthetic requirements, hemodynamic parameters, and adverse events during non-intubated VATS.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) score of I-III patients receiving video-assisted thoracoscopic surgery

Exclusion Criteria:

* Age < 18 or > 80 years
* ASA classifications > III
* Pregnancy
* Known allergies to any drugs used in the study
* Emergency surgery
* Patient refusal
* Chronic pain history

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Cough | Intraoperative period
  The incidence of cough reflex during surgery and severity Cough severity: 1=none, 2=slight, 3=moderate, 4=severe

SECONDARY OUTCOMES:
Intraoperative fentanyl consumption | Intraoperative period
  Fentanyl bolus for cough reflex and limb movement
Total fentanyl consumption | Intraoperative period
  Total fentanyl requirement during surgery
Total propofol consumption | Intraoperative period
  Total propofol requirement during surgery
Intraoperative adverse events | Intraoperative period
  The incidence of hypotension, bradycardia and hypoxia
Postoperative numeric rating scale | Postoperative 48 hours
  Numeric rating scale within postoperative 48 hours NRS scores is labeled from zero to ten, with zero being an example of someone with no pain and ten being the worst pain possible.
Postoperative opioid requirement | Postoperative 48 hours
  Postoperative opioid requirement within postoperative 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
There is no plan to share

REFERENCES:
- [Background] Feray S, Lubach J, Joshi GP, Bonnet F, Van de Velde M; PROSPECT Working Group *of the European Society of Regional Anaesthesia and Pain Therapy. PROSPECT guidelines for video-assisted thoracoscopic surgery: a systematic review and procedure-specific postoperative pain management recommendations. Anaesthesia. 2022 Mar;77(3):311-325. doi: 10.1111/anae.15609. Epub 2021 Nov 5. PMID 34739134
- [Background] Selim J, Jarlier X, Clavier T, Boujibar F, Dusseaux MM, Thill J, Borderelle C, Ple V, Baste JM, Besnier E, Djerada Z, Compere V. Impact of Opioid-free Anesthesia After Video-assisted Thoracic Surgery: A Propensity Score Study. Ann Thorac Surg. 2022 Jul;114(1):218-224. doi: 10.1016/j.athoracsur.2021.09.014. Epub 2021 Oct 15. PMID 34662540
- [Background] Wang YL, Kong XQ, Ji FH. Effect of dexmedetomidine on intraoperative Surgical Pleth Index in patients undergoing video-assisted thoracoscopic lung lobectomy. J Cardiothorac Surg. 2020 Oct 2;15(1):296. doi: 10.1186/s13019-020-01346-1. PMID 33008451
- [Background] Wang XR, Jia XY, Jiang YY, Li ZP, Zhou QH. Opioid-free anesthesia for postoperative recovery after video-assisted thoracic surgery: A prospective, randomized controlled trial. Front Surg. 2023 Jan 6;9:1035972. doi: 10.3389/fsurg.2022.1035972. eCollection 2022. PMID 36684254
- [Background] Lee SH, Lee CY, Lee JG, Kim N, Lee HM, Oh YJ. Intraoperative Dexmedetomidine Improves the Quality of Recovery and Postoperative Pulmonary Function in Patients Undergoing Video-assisted Thoracoscopic Surgery: A CONSORT-Prospective, Randomized, Controlled Trial. Medicine (Baltimore). 2016 Feb;95(7):e2854. doi: 10.1097/MD.0000000000002854. PMID 26886651